CLINICAL TRIAL: NCT02760056
Title: Thyroid Hormone for Remyelination in Multiple Sclerosis (MS): A Safety and Dose Finding Study
Acronym: MST3K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michelle Cameron, Chair and Roy & Eulalia Swank Family Research Professor, Oregon Health and Science University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 15101
Record Dates: First submitted 2016-04-05; First posted 2016-05-03 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: Thyroid hormone; Remyelination
MeSH Terms: conditions — Multiple Sclerosis | interventions — Triiodothyronine

STUDY DESIGN:
Intervention Model Description: Dose escalation with monitoring for safety and tolerability, as well as reliability of VEP testing.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, randomized, controlled
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liothyronine (cytomel) (Active Comparator): Subjects will be divided into 4 groups. The first group will take 25 mcg twice daily for one week. The second group will take 37.5 mcg twice daily for one week. The third group will take 50 mcg twice daily for one week. The firth group will take 75 mcg twice daily for one week
  Interventions: Drug: Liothyronine sodium
- Placebo (Placebo Comparator): Subject will take matching placebo twice a day for one week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liothyronine sodium — Subjects will be divided into 4 groups of progressively escalating doses. Each group will have 6 subjects 4 will receive the active treatment and 2 will receive the placebo. The first group will receive 25 mcg twice daily for one week. The second group will receive 37.5 mcg twice daily for one week. The third group will receive 50 mcg twice daily for one week. The forth group will receive 75 mcg twice daily for one week.
  Other Names: Cytomel
  Arms: Liothyronine (cytomel)
Drug: Placebo — Patient will receive a matching placebo to take twice daily for one week.
  Arms: Placebo

SUMMARY:
This is a phase 1 study evaluating the safety and maximum tolerated dose of Liothyronine (T3) in subjects with multiple sclerosis

DETAILED DESCRIPTION:
This is a pilot, phase I, placebo controlled clinical trial of short-term high-dose thyroid hormone to promote remyelination in MS. Permanent clinical disability in MS is likely caused by the neuronal damage and degeneration that follows recurrent demyelination with progressive failure of remyelination. Thyroid hormone (TH) is required for central nervous system (CNS) myelination during development, and CNS remyelination in animal models of MS, a process similar to developmental myelination, has also been found to be promoted by TH. This study will ascertain the safety, tolerability and maximum tolerated dose of TH in people with MS, explore reliability for a potential signal of treatment efficacy and mechanism, and optimize procedures for a full scale clinical trial to evaluate the efficacy of pulsed TH for promotion of remyelination in MS.

The safety and tolerability of this treatment will be assessed using subjects' self-report of symptoms, the validated Hyperthyroid Symptom Scale (HSS), and blood pressure measurements. a

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS of any type
* Age 18 to 50 years
* Weight range 45-90 kg (100-200 lbs)
* Lesions on brain MRI

Exclusion Criteria:

* History of hypo or hyperthyroidism and a normal TSH
* History of high blood pressure (hypertension) [
* Resting blood pressure greater than 150/95, resting heart rate greater than 100
* History of coronary artery disease or clinically significant arrhythmia, clinically significant abnormalities on EKG
* History of diabetes
* History of anemia or renal (kidney) disease
* Clinically significant abnormalities on metabolic panel or serum hematocrit below 32 %
* History of atrophic gastritis
* History of anxiety disorder or bipolar disorder
* Serious psychiatric or medical conditions that would preclude reliable participation in the study
* Use of illicit substances or alcohol abuse
* Current use of fingolimod (Gilenya)
* Current or prior use of mitoxantrone (Novantrone)
* Current use of stimulants (methylphenidate, atomoxetine, dextroamphetamine,phentermine)
* Current use of any blood thinners such as warfarin or apixaban (Aspirin is ok)
* Medications which would metabolized faster in the presence of thyroid hormone (Insulin, oral hypoglycemic agents and oral anticoagulants)
* Severe head tremors (which would impair the ability to perform VEPs)
* Present or recent use of medications that could interact with the thyroid hormone (iodine containing agents such as kelp supplements, amiodarone, iodinated contrast given for CT or xray), P450 stimulants (phenytoin, carbamazepine, phenobarbital, and rifampin)
* Corrected visual acuity worse than 20/50 in either eye or other eye issues that would prevent reading of a standard eye chart
* Head tremors or other tremors that would prevent sitting relatively still for a vision test
* Patients taking proton pump inhibitors (PPIs) or H2 blockers will be excluded unless they can safely not take these medications during the week of study drug administration.
* Patients taking Ampyra (dalfampridine) will be excluded unless they can safely not take these medications during the week of study drug administration.
* Pregnancy, breastfeeding, or intention to become pregnant in the following month
* Inability to receive an MRI (e.g. implanted metal device)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cameron, MD, Principal Investigator — OHSU Department of Neurology
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wooliscroft L, Altowaijri G, Hildebrand A, Samuels M, Oken B, Bourdette D, Cameron M. Phase I randomized trial of liothyronine for remyelination in multiple sclerosis: A dose-ranging study with assessment of reliability of visual outcomes. Mult Scler Relat Disord. 2020 Jun;41:102015. doi: 10.1016/j.msard.2020.102015. Epub 2020 Feb 20. PMID 32120028

RESULTS

PARTICIPANT FLOW:
Groups:
- Liothyronine (Cytomel): Subjects will be divided into 4 groups. The first group will take 25 mcg twice daily for one week. The second group will take 37.5 mcg twice daily for one week. The third group will take 50 mcg twice daily for one week. The firth group will take 75 mcg twice daily for one week
  Liothyronine sodium: Subjects will be divided into 4 groups of progressively escalating doses. If the study is fully enrolled, each group will have 6 subjects 4 will receive the active treatment and 2 will receive the placebo. The first group will receive 25 mcg twice daily for one week. The second group will receive 37.5 mcg twice daily for one week. The third group will receive 50 mcg twice daily for one week. The forth group will receive 75 mcg twice daily for one week.
Period: Overall Study
Arm/Group | Liothyronine (Cytomel) | Placebo
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liothyronine (Cytomel) | Placebo | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Full Range); unit: years] | 39 [30 to 49] | 38.4 [21 to 46] | 38.8 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 4 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
MS Subtype [Count of Participants; unit: Participants]
  Relapsing Remitting Multiple Sclerosis | 9 | 5 | 14
  Secondary Progressive Multiple Sclerosis | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) of Oral L-T3 in Subjects With MS
Description: MTD per protocol (dose level one category below dose at which study was stopped due to intolerance or meeting criteria for cessation)
Time Frame: 1 week
Population: Participants with MS taking L-T3 (10) excluding those taking placebo (5)
Measure: Number; unit: mcg daily with BID dosing
Arm/Group | Liothyronine (Cytomel)
Number analyzed (Participants) | 10
mcg daily with BID dosing | 75

2. Secondary Outcome: Reliability of Visual Evoked Potential (VEP) Testing (ICC)
Description: P100 latency will be compared before and after treatment with L-T3 in subjects receiving the active treatment to assess reliability of the test for future assessment of treatment effect.
Time Frame: 1 week
Population: Participants with MS taking L-T3 or placebo
Measure: Number; unit: Intraclass Coefficient (ICC)
Groups:
- All Participants: Measure value across cohorts.
Arm/Group | Liothyronine (Cytomel) | Placebo | All Participants
Number analyzed (Participants) | 10 | 5 | 15
Intraclass Coefficient (ICC)
  ICC - Right Eye | 0.852 | 0.679 | 0.824
  ICC - Left Eye | 0.746 | 0.966 | 0.845
  ICC- Mixed Model | 0.889 | 0.963 | 0.924

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Liothyronine (Cytomel) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 6/10 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (Cytomel) (N=10) | Placebo (N=5)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Poor Sleep (Psychiatric disorders) | 4 | 1
Loose Stool (Gastrointestinal disorders) | 5 (5) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (7)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Back and Leg pain
Yellow stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased severity in post-Tecfidera flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Self-reporting of BP, HR. 1 missed dose in the drug arm. VEP testing was conducted by multiple technicians and read by multiple attending physicians; though visit one and two were more often conducted by the same tech/attending.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes